CLINICAL TRIAL: NCT06052007
Title: In-Situ Simulation Study Among Nurses Using Different Debriefing Methods
Brief Title: In-Situ Simulation Different Debriefing Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, özlem doğu, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Different Debriefing Methods
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Nursing Caries; Satisfaction; Simulation of Physical Illness
Keywords: in-situ simulation; critical thinking; debriefing; nurse; intensive care
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LC-Based Debriefing (Experimental): LC-based debriefing session in one intervention group.
  Interventions: Behavioral: LC-Based Debriefing
- 3D Model-Based Debriefing (Experimental): One facilitator conducted a 3D model-based debriefing session in the other intervention group.
  Interventions: Behavioral: 3D Model-Based Debriefing
- Standard Debriefing (No Intervention): One facilitator conducted a non-model-based unstructured debriefing session in the control group

INTERVENTIONS:
Behavioral: LC-Based Debriefing — LC-based debriefing encourages reflection by allowing learners to identify and explore topics of particular interest. The model is defined as a structured post-event LC, which is useful for improving competence, professional development, and clinical judgment among intensive care unit and trauma nurses. The model is useful not only for one recipient by allowing reflection on positive and negative experiences but also for the whole group by allowing them to make connections to their own practice that day or to previous experiences, supporting teamwork. It also helps them understand what good practice is by doing their own self-assessment with peers' benchmarking.
  Arms: LC-Based Debriefing
Behavioral: 3D Model-Based Debriefing — The model has three parts: defusing, discovering, and deepening. The experiential learning theory on which this model is based facilitates learning goals. This model allows its participants to create new mental models for future practice, develop critical thinking skills, and identify knowledge gaps. In the model, a debriefing session starts with preliminary information and ends with a summary of what has been learned. Participants' gaps in understanding and learning are identified, and how they can apply their learnings to practice is discussed.
  Arms: 3D Model-Based Debriefing

SUMMARY:
The goal of this pre-test-post-test randomized controlled experimental study is to examined the effects of the learning conversation (LC)-based, 3D model-based, and standard debriefing methods on critical thinking, debriefing experience, and satisfaction after in-situ simulation among intensive care unit (ICU) nurses.

A total of 186 ICU nurses working in a training and research hospital participated in the study. Researchers will compare learning conversation (LC)-based, 3D model-based, and standard debriefing methods on critical thinking, debriefing experience, and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Volunterring
* Beclohers degree graduated
* 22- 55 years
* min 1 year to work as a nurse
* open to communication

Exclusion Criteria:

* individuals outside the inclusion criteria

Ages: 23 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Examined criticical thinking knownledge test score of intervention and control groups | 2 months
  The criticical thinking knownledge test was also created by the researchers and comprised 10 questions about learning objectives and critical thinking, particularly regarding decision-making while performing elimination, nutritional, and respiratory activities of ICU patients.
Determinating satisfaction scores of intervention and control groups | 2 months
  A visual analog scale (0 = not at all satisfied, 10 = very satisfied), the participants were asked to rate their satisfaction.
Determinating debriefing experince score of intervention and control groups | 2 months
  The Debriefing Experience Scale consists of 20 items and is a 5-point Likert-type scale. It consists of two parts-experience with debriefing and importance of items-and four subscales-analyzing thoughts and feelings, learning and making connections, facilitator skill in conducting the debriefing, and appropriate facilitator guidance. A high score on the scale indicates increased gains from the debriefing experience

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data set can be shared
Supporting Information: SAP

REFERENCES:
- [Result] Abu-Sultaneh S, Whitfill T, Rowan CM, Friedman ML, Pearson KJ, Berrens ZJ, Lutfi R, Auerbach MA, Abulebda K. Improving Simulated Pediatric Airway Management in Community Emergency Departments Using a Collaborative Program With a Pediatric Academic Medical Center. Respir Care. 2019 Sep;64(9):1073-1081. doi: 10.4187/respcare.06750. Epub 2019 Apr 23. PMID 31015388
- [Result] Almomani E, Sullivan J, Hijjeh M, Attlallah K. The perceived relationship between reflective learning conversation and clinical reasoning skills amongst critical care and trauma nurses: A cross sectional parallel mixed method. Nurse Educ Today. 2021 Oct;105:105044. doi: 10.1016/j.nedt.2021.105044. Epub 2021 Jul 2. PMID 34242908
- [Result] Baldwin LJ, Jones CM, Hulme J, Owen A. Use of the learning conversation improves instructor confidence in life support training: An open randomised controlled cross-over trial comparing teaching feedback mechanisms. Resuscitation. 2015 Nov;96:199-207. doi: 10.1016/j.resuscitation.2015.08.010. Epub 2015 Aug 24. PMID 26316279
- [Result] Dochez V, Beringue F, Legendre G, Jeanneteau P, Rolland D, Coutin AS, Collin R, Boulvais E, Malo L, Chupin AM, Cousin B, Flamant C, Winer N. Assessment of a multiprofessional training programme by in situ simulation in the maternity units of the Pays de Loire regional perinatal network. J Gynecol Obstet Hum Reprod. 2021 Sep;50(7):102107. doi: 10.1016/j.jogoh.2021.102107. Epub 2021 Mar 8. PMID 33705991
- [Result] Kang K, Yu M. Comparison of student self-debriefing versus instructor debriefing in nursing simulation: A quasi-experimental study. Nurse Educ Today. 2018 Jun;65:67-73. doi: 10.1016/j.nedt.2018.02.030. Epub 2018 Mar 2. PMID 29533836
- [Result] Lee J, Lee H, Kim S, Choi M, Ko IS, Bae J, Kim SH. Debriefing methods and learning outcomes in simulation nursing education: A systematic review and meta-analysis. Nurse Educ Today. 2020 Apr;87:104345. doi: 10.1016/j.nedt.2020.104345. Epub 2020 Jan 16. PMID 32135455
- [Result] Niu Y, Liu T, Li K, Sun M, Sun Y, Wang X, Yang X. Effectiveness of simulation debriefing methods in nursing education: A systematic review and meta-analysis. Nurse Educ Today. 2021 Dec;107:105113. doi: 10.1016/j.nedt.2021.105113. Epub 2021 Aug 27. PMID 34492539
- [Result] Reed SJ. Written debriefing: Evaluating the impact of the addition of a written component when debriefing simulations. Nurse Educ Pract. 2015 Nov;15(6):543-8. doi: 10.1016/j.nepr.2015.07.011. Epub 2015 Aug 5. PMID 26299701
- [Result] Villemure C, Georgescu LM, Tanoubi I, Dube JN, Chiocchio F, Houle J. Examining perceptions from in situ simulation-based training on interprofessional collaboration during crisis event management in post-anesthesia care. J Interprof Care. 2019 Mar-Apr;33(2):182-189. doi: 10.1080/13561820.2018.1538103. Epub 2018 Nov 5. PMID 30395755